CLINICAL TRIAL: NCT06158113
Title: Efficacy and Safety of Baricitinib for the Treatment of Oral Lichen Planus: A Proof-of-Concept Study
Brief Title: Efficacy and Safety of Baricitinib in Oral Lichen Planus: a Proof-of-Concept Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-0969
Record Dates: First submitted 2023-11-27; First posted 2023-12-06 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Lichen Planus, Oral; Lichen Planus, Mucosal; Oral Lichen Planus
Keywords: Jak inhibitor; Janus kinase inhibitor
MeSH Terms: conditions — Lichen Planus, Oral; Lichen Planus | interventions — baricitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Baricitinib (Experimental): Participants will be asked to take 4mg of baricitinib by mouth daily for up to 24 weeks.
  Interventions: Drug: Baricitinib 4 milligram Oral Tablet

INTERVENTIONS:
Drug: Baricitinib 4 milligram Oral Tablet — 4 milligrams once daily
  Other Names: Olumiant

SUMMARY:
The goal of this clinical trial is to learn the effects of baricitinib (the study drug) in patients with Oral Lichen Planus. The main questions it aims to answer are:

* What is the efficacy of baricitinib in treating moderate to severe Oral Lichen Planus?
* Can baricitinib treatment in Oral Lichen Planus change quality of life?
* What side effects do patients with Oral Lichen Planus experience when treated with baricitinib?

Participants will be required to come in to monthly visits for up to eight months. During visits, participants will be:

* Evaluated for the extent of their disease
* Asked to fill out a questionnaire about their quality of life
* Given baricitinib for them to take at home for six months
* Evaluated for any potential side experienced while on treatment
* Asked to return 1 month after completing treatment

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signed an Institutional Review Board (IRB) approved informed consent.
2. Be at least ≥ 18 years old.
3. Biopsy proven Oral Lichen Planus (OLP)
4. OLP patients with moderate to severe OLP, and must have failed or not tolerated at least one non-corticosteroid systemic treatment for OLP (such as metronidazole, hydroxychloroquine, methotrexate, mycophenolate mofetil, azathioprine, acitretin, rituximab, thalidomide, cyclosporine, apremilast, dapsone or systemic calcineurin inhibitor).
5. Subjects should practice daily oral hygiene (defined as brushing teeth twice daily) and be willing to maintain their routine oral hygiene procedure during study participation.
6. Willingness to abstain from certain mouth products during the course of the study
7. Must be willing to not receive any live vaccines during and up to 30 days after the end of treatment.
8. Vaccination status of subjects should be reviewed prior to study entry. Subjects must be encouraged to receive non-live vaccines following centers of disease control (CDC) guidelines for vaccination of those ≥18 years of age to prevent infectious disease 30 days before baseline.
9. Individuals who can potentially become pregnant must have a negative urine pregnancy test at screening and must be confirmed negative at time of enrollment (baseline visit).
10. Individuals who can potentially become pregnant must agree to use a highly effective form of birth control when engaging in sexual intercourse with a male partner during the study and for 30 days after the last dose.
11. Male subjects must be willing to use a highly effective method of contraception or practice true abstinence from sexual intercourse during the study and for 30 days after the last dose.
12. Must be able to comply with study instructions and attend all study visits.

Exclusion Criteria:

1. Absolute lymphocyte count <750cells/mm^3 within 30 days of starting study drug
2. Absolute neutrophil count <1200cells/mm^3 within 30 days of starting study drug
3. Hemoglobin <10.0g/dL within 30 days of starting study drug
4. Platelet count <100,000 cells/mm^3 within 30 days of starting study drug
5. Fasting cholesterol levels >400mg/dL or >10.34mmol/L within 30 days of starting study drug or levels that may have required hospitalization, caused pancreatitis, or became life threatening.
6. Serum triglycerides >500mg/dL or >5.7mmol/L within 30 days of starting study drug.
7. Chronic liver disease with severe hepatic impairment as defined in the protocol.
8. Inadequate renal function tests defined as an estimated glomerular filtration rate (eGFR) based on the most recent available creatinine using the chronic kidney disease epidemiology collaboration equation (CKD-EPI) creatinine 2009 equation of <60 millimeters/minute/1.73 meters squared (m^2) within 30 days of starting study drug.
9. Ongoing active or recent clinically serious fungal, bacterial, viral, or parasitic infection.
10. History of gastrointestinal perforation
11. History of heart attack or significant cardiovascular risk that in the investigator's judgement, the risks of the subject participating in the study is greater than its benefit.
12. Hypercoagulable state such as history of deep vein thromboembolism (VTE) or stroke OR are considered at high risk of VTE.
13. History of cancer (except treated cutaneous basal cell carcinoma (BCC), cutaneous squamous cell carcinoma in situ (cSCCis) and in situ cervical cancer) unless it can be documented that the patient has been in a disease-free state for at least 5 years for high grade cancers with the following exception:

    * In case of clinical suspicion of malignancy in the oral cavity, a patient can only be included after an excluding biopsy
    * Any history of squamous cell carcinoma or melanoma (even if resected) in the mouth, as well as history of other non-squamous cell carcinoma (e.g., sarcoma, salivary gland tumors) in the mouth are excluded.
14. Subjects who may have signs of lymphoproliferative disease, such as lymphadenopathy or splenomegaly unless stable for the last 5 years
15. Professional dental cleaning within 2 weeks prior to baseline
16. Patient with any un-healed oral surgery (including recent diagnostic biopsies, if applicable) or oral laser therapeutic wound(s) at baseline visit
17. Subjects must have failed at least one systemic therapy for OLP to be included in the study. Appropriate washout for past medications received and stable doses for other medications should be followed as outlined in the protocol.
18. Hypersensitivity to Janus kinase (JAK) inhibitors.
19. Subjects with any serious concomitant illness that is anticipated to require the use of systemic corticosteroids or otherwise interfere with study participation or require active frequent monitoring (e.g., unstable chronic asthma)
20. Subjects who require major surgery within 8 weeks of baseline and/or during the study are excluded.
21. Current participation in another clinical study and/or having received treatment with any non-marketed / investigational medicinal product (drug substance or medical device) within 30 days prior to baseline or 5.5 half-lives, whichever is longer.
22. Intention to become pregnant during the study period (30 days after stopping investigational product)
23. Intention to breastfeed until 30 days after stopping investigational product.
24. Any other condition that in the investigator's judgement the subject's risks are greater than the benefit from participating in the study or may interfere with interpretation of data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in Oral Disease Severity Scale (ODSS) Scores | Baseline, 24 weeks
  The Oral Disease Severity Scale (ODSS) is a validated tool to assess severity of Oral Lichen Planus. For scoring, the oral cavity is divided into 17 sites and assigned three different scores. A site score, which captures disease extent, a severity score, and an activity score which is obtained by multiplying the site and severity scores. Independently study participants are asked to fill in a numerical rating scale graded from 0-10, with zero meaning no pain and 10 being the worst imaginable pain felt within the last 4 weeks. Scores are added together and range from 0-106, with higher scores meaning more severe disease. Overall change from baseline to week 24 will be reported.

SECONDARY OUTCOMES:
Changes in Quality of Life as assessed with the Chronic Oral Mucosal Disease Questionnaire-26 (COMDQ-26). | Baseline, 24 weeks
  The Chronic Oral Mucosal Disease Questionnaire-26 (COMDQ-26) is a 26-item validated survey specific to assess changes in quality of life in patients with Oral Lichen Planus. The total score of the COMDQ-26 ranges from 0-104 with higher scores indicating worse quality of life. The number of participants that achieve at least a 9 point reduction in their scores from baseline will be reported.

OTHER OUTCOMES:
Estimated response to 24 weeks of treatment with 4mg of baricitinib daily using the Investigator's Global Assessment (IGA). | Baseline, 24 weeks
  The Investigator Global Assessment (IGA) represents the study doctor's overall assessment of the extent of disease. It assesses changes in symptomatic Oral Lichen Planus and it is meant to be a well-defined and reliable tool to measure disease severity in clinical studies. This tool assigns a score of 0-4 depending on how severe the disease is, with higher scores meaning worse disease. Overall change from baseline to week 24 reported.

CONTACTS AND LOCATIONS:
Overall Officials: Donna Culton, MD, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Dermatology and Skin Cancer Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University of North Carolina at Chapel Hill.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 and continuing for 36 months after publication.
Access Criteria: Data will be made available to investigators who have approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University of North Carolina at Chapel Hill.

REFERENCES:
- [Background] Escudier M, Ahmed N, Shirlaw P, Setterfield J, Tappuni A, Black MM, Challacombe SJ. A scoring system for mucosal disease severity with special reference to oral lichen planus. Br J Dermatol. 2007 Oct;157(4):765-70. doi: 10.1111/j.1365-2133.2007.08106.x. Epub 2007 Aug 17. PMID 17711534
- [Background] Wiriyakijja P, Porter S, Fedele S, Hodgson T, McMillan R, Shephard M, Ni Riordain R. Meaningful improvement thresholds in measures of pain and quality of life in oral lichen planus. Oral Dis. 2020 Oct;26(7):1464-1473. doi: 10.1111/odi.13379. Epub 2020 May 26. PMID 32363637
- [Background] Damsky W, Wang A, Olamiju B, Peterson D, Galan A, King B. Treatment of severe lichen planus with the JAK inhibitor tofacitinib. J Allergy Clin Immunol. 2020 Jun;145(6):1708-1710.e2. doi: 10.1016/j.jaci.2020.01.031. Epub 2020 Feb 1. No abstract available. PMID 32018031
- [Background] Shao S, Tsoi LC, Sarkar MK, Xing X, Xue K, Uppala R, Berthier CC, Zeng C, Patrick M, Billi AC, Fullmer J, Beamer MA, Perez-White B, Getsios S, Schuler A, Voorhees JJ, Choi S, Harms P, Kahlenberg JM, Gudjonsson JE. IFN-gamma enhances cell-mediated cytotoxicity against keratinocytes via JAK2/STAT1 in lichen planus. Sci Transl Med. 2019 Sep 25;11(511):eaav7561. doi: 10.1126/scitranslmed.aav7561. PMID 31554739